CLINICAL TRIAL: NCT06638957
Title: Impact of the Coronavirus Disease 2019 Pandemic on Oncologic Outcomes in Colorectal Cancer
Brief Title: Impact of the COVID-19 Pandemic on Oncologic Outcomes in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: In Ja Park (Other)
Collaborators: Kyungpook National University Chilgok Hospital (Other); Gangnam Severance Hospital (Other); Chonnam National University Hospital (Other); Korea University Anam Hospital (Other); Pusan National University Yangsan Hospital (Other); Samsung Medical Center (Other); Seoul Saint Mary's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, In Ja Park, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: COVID
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Carcinoma; COVID 19
Keywords: colorectal; covid; oncologic outcome
MeSH Terms: conditions — Colorectal Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with colorectal cancer who underwent surgical treatment from 2018 to 2020: The pre-COVID-19 period extended from 2018 to February 2020
- patients with colorectal cancer who underwent surgical treatment from 2020: the COVID-19 period began in March 2020 to December 2020

SUMMARY:
The goal of this observational study is to assess the impact of the COVID-19 pandemic on colorectal cancer (CRC) outcomes, particularly focusing on stage distribution and recurrence-free survival in patients undergoing surgery at eight tertiary care institutions in Korea from 2018 to 2020.

Main Question Does the COVID-19 pandemic lead to more advanced stages of colorectal cancer at diagnosis and higher complication rates during surgery? Is there a significant difference in recurrence-free survival between CRC patients treated before and during the pandemic?

This study found that more patients presented with advanced-stage CRC during the COVID-19 pandemic, with significantly higher rates of tumor-related complications (perforations, abscesses, and preoperative obstructions), as well as an increase in open surgeries and combined resections.

No significant difference in recurrence-free survival was observed between the pre-COVID-19 and COVID-19 periods, although postoperative complication rates were higher, especially among rectal cancer patients and those receiving preoperative chemoradiotherapy.

DETAILED DESCRIPTION:
This observational, population-based, cohort study was conducted in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology guidelines. It was approved by the regional ethics committee in the Republic of Korea and institutional review boards of the eight participating institutions. Due to the anonymity of the data, the requirement for informed consent was waived.

The study timeline was determined by the phased social distancing measures implemented in the Republic of Korea in response to the COVID-19 pandemic. The study focused on patients with CRC who underwent surgical treatment from 2018 to 2020. The pre-COVID-19 period extended from 2018 to February 2020, and the COVID-19 period began in March 2020 with the identification of the first COVID-19 case in the Republic of Korea and subsequent government measures to prevent the spread of the disease.

Eight institutions across the Republic of Korea participated in the study, including Asan Medical Center, Seoul St. Mary's Hospital, Korea University Anam Hospital, Samsung Medical Center, Pusan National University Yangsan Hospital, Gangnam Severance Hospital, Kyungpook National University Chilgok Hospital, and Chonnam National University Hwasun Hospital. These institutions are tertiary medical centers, varying in location and size.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal cancer who underwent surgery
* in 8 institution including Asan Medical Center, Seoul St. Mary's Hospital, Korea University Anam Hospital, Samsung Medical Center, Pusan National University Yangsan Hospital, Gangnam Severance Hospital, Kyungpook National University Chilgok Hospital, and Chonnam National University Hwasun Hospital

Exclusion Criteria:

* Familial adenomatous polyposis (FAP)
* Hereditary non-polyposis colon cancer (HNPCC)
* Cancer associated with inflammatory bowel disease (IBD)
* Colorectal cancer not proven on biopsy, and pathologies other than adenocarcinoma.
* Emergency operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between 2018 and 2020, 14951 patients underwent surgery for suspected CRC across the eight institutions.
Sampling Method: Non-Probability Sample
Enrollment: 14951 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
stage distribution in patients who underwent CRC surgery during the pre-COVID-19 period, compared with those who underwent the surgery during the COVID-19 period. | At the time the biopsy results were available for patients who underwent surgery between 2018 and 2020 (7 days after surgery).
  We aimed to document the pathological stage for each patient based on the biopsy results after surgery and analyze how the stage distribution differed between the pre-COVID and COVID groups.

SECONDARY OUTCOMES:
2-year recurrence free survival (RFS) and surgical complication rate in patients who underwent CRC surgery during the pre-COVID-19 period, compared with those who underwent the surgery during the COVID-19 period. | Outcome measures will be assessed at 2 years post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No